CLINICAL TRIAL: NCT05760547
Title: The Translational Initiative to Map Epigenetics in Aging (TIME-A)
Acronym: TIME-A
Status: Not yet recruiting | Type: Observational
Sponsor: Elysium Health (Industry)
Responsible Party: Sponsor
Other Study IDs: TIME-A
Record Dates: First submitted 2023-02-09; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Biological Aging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIME-A: Group will complete periodic surveys

SUMMARY:
The Translational Initiative to Map Epigenetics in Aging (TIME-A) study aims to advance our understanding of the connections between epigenetics, lifestyle, demographics, and health and aging.

DETAILED DESCRIPTION:
TIME-A is a longitudinal research initiative. Anyone who has ever taken an Index test registered through Elysium Health is eligible to participate. Participation involves answering questions that will be administered via a survey format. Research participants' survey responses will be combined with their epigenetic Index data with the primary aim of identifying the contributions of 1) environmental and lifestyle factors, 2) general health, and 3) medical history, on biological age. Exploratory aims include the development of epigenetic signatures that are predictive of health status, and exploring the relationship between epigenetically-derived health phenotypes and biological age. These findings will lay the foundation for personalized health recommendations using Index (including, but not limited to: workout routines, diets, supplement regimens, medications, lifestyle changes).

ELIGIBILITY:
Inclusion Criteria:

* All adults aged 18 and above
* Have registered at least one Index kit via the Elysium Health website
* Able and willing to provide digital consent to the Research Consent Form, and the TIME-A Research Subject Consent Form

Exclusion Criteria:

* Consent to participate not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 or older
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2023-03-08 (Estimated); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of environmental and lifestyle factors on biological age | At baseline and throughout study (approximately every 6 months up to 120 months)
  Univariate and multivariate statistical methods will be used to identify which environmental and lifestyle factors (from TIME-A survey responses) influence biological age.
Effect of general health on biological age | At baseline and throughout study (approximately every 6 months up to 120 months)
  Univariate and multivariate statistical methods will be used to identify which general health characteristics (from TIME-A survey responses) influence biological age.
Effect of medical history on biological age | At baseline and throughout study (approximately every 6 months up to 120 months)
  Univariate and multivariate statistical methods will be used to identify the impact of medical history (from TIME-A survey responses) on biological age.

OTHER OUTCOMES:
Develop epigenetic signatures that are predictive of health status | At baseline and throughout study (approximately every 6 months up to 120 months)
  DNA methylation data and TIME-A survey responses will be combined. Supervised and unsupervised machine learning methods will be used to generate novel methylation-derived predictors of participants' survey responses.

CONTACTS AND LOCATIONS:
Overall Officials: Dayle Sampson, PhD, Principal Investigator — Elysium Health; Holly Holmes, PhD, Principal Investigator — Elysium Health

IPD SHARING:
Plan to Share IPD: No